CLINICAL TRIAL: NCT05179239
Title: A Randomized，Double-blind，Controlled，Multi-center Phase III Clinical Study Evaluating SHR-1701 or Placebo Plus Chemotherapy With or Without BP102 (Bevacizumab) as First-Line Treatment in Patients With Persistent, Recurrent, or Metastatic Cervical Cancer
Brief Title: A Study of SHR-1701 Plus Platinum-containing Chemotherapy With or Without BP102 (Bevacizumab) as First-line Treatment in Cervical Cancer
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor develops strategy adjustment
Sponsor: Suzhou Suncadia Biopharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHR-1701-III-309
Record Dates: First submitted 2021-10-14; First posted 2022-01-05 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — SHR-1701; Paclitaxel; Cisplatin; Carboplatin

STUDY DESIGN:
Intervention Model Description: SHR-1701 or Placebo Plus Chemotherapy With or Without BP102 (Bevacizumab)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SHR-1701 + paclitaxel + cisplatin/carboplatin + BP102 (Experimental)
  Interventions: Drug: SHR-1701 + paclitaxel + cisplatin/carboplatin + BP102
- SHR-1701 + paclitaxel + cisplatin/carboplatin ± BP102 (Experimental)
  Interventions: Drug: SHR-1701 + paclitaxel + cisplatin/carboplatin± BP102
- Placebo + paclitaxel + cisplatin/carboplatin ± BP102 (Placebo Comparator)
  Interventions: Drug: Placebo + paclitaxel + cisplatin/carboplatin ± BP102

INTERVENTIONS:
Drug: SHR-1701 + paclitaxel + cisplatin/carboplatin + BP102 — SHR-1701 + paclitaxel + cisplatin/carboplatin + BP102
  Arms: SHR-1701 + paclitaxel + cisplatin/carboplatin + BP102
Drug: SHR-1701 + paclitaxel + cisplatin/carboplatin± BP102 — SHR-1701 + paclitaxel + cisplatin/carboplatin± BP102
  Arms: SHR-1701 + paclitaxel + cisplatin/carboplatin ± BP102
Drug: Placebo + paclitaxel + cisplatin/carboplatin ± BP102 — Placebo + paclitaxel + cisplatin/carboplatin ± BP102
  Arms: Placebo + paclitaxel + cisplatin/carboplatin ± BP102

SUMMARY:
The study is being conducted to evaluate the efficacy, and safety of SHR-1701 or Placebo Plus Chemotherapy With or Without BP102 (Bevacizumab) as First-Line Treatment in Patients With Persistent, Recurrent, or Metastatic Cervical Cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-70 years, female.
2. With Eastern Cooperative Oncology Group (ECOG) performance status scores of 0-1.
3. With a life expectancy of ≥ 12 weeks.
4. Acute toxicities from prior anti-tumor treatments must have resolved to Grade 0-1 (per NCI CTCAE 5.0).
5. With at least one measurable lesion as per RECIST v1.1.
6. With histologically confirmed squamous cell carcinoma, adenocarcinoma, or adenosquamous cell carcinoma of the cervix.
7. Persistent, recurrent, or metastatic cervical cancer.
8. Patients to be enrolled in Stage II are required to provide a minimum of 10 slides of fresh (preferred).
9. Women of childbearing potential must have a negative serum pregnancy test within 3 days prior to starting study treatment.
10. Patients must agree and have signed the informed consent form.

Exclusion Criteria:

1. With known contraindications to paclitaxel, cisplatin, or carboplatin.
2. With known allergies to any of the study drugs or their excipients; severe allergic reactions to other monoclonal antibodies.
3. With inadequately treated CNS metastasis.
4. With uncontrolled hypertension.
5. With uncontrolled cardiac diseases or symptoms.
6. With major vascular disease.
7. With arterial/venous thrombotic events within 6 months prior to randomization.
8. Have received full-dose anticoagulant or hemolytic therapy within 10 days prior to randomization.
9. With clinically significant hemorrhage or definitive bleeding diathesis within 3 months prior to randomization.
10. With severe, unhealed, or open wounds as well as active ulcers or untreated fractures.
11. With any active autoimmune disease or a history of autoimmune disease that is expected to recur.
12. Had other active malignant tumors within 5 years prior to study enrolment.
13. With congenital or acquired immunodeficiency (such as HIV-infected patients).

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2022-02-26 (Actual); Primary Completion 2024-08-12 (Actual); Study Completion 2024-08-12 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of Participants Who Experience an Adverse Event (AE) as per NCI-CTC AE 5.0（Stage I） | Up to approximately 21 days
Incidence and severity of Participants Who Experience a Serious AE (SAE) as per NCI-CTC AE 5.0（Stage I） | Up to approximately 21 days
Incidence and severity of Participants Who Experience an Immune-related AE (irAE) as per NCI-CTC AE 5.0（Stage I） | Up to approximately 21 days
BIRC-assessed progression-free survival (PFS) as per RECIST v1.1（Stage II） | Up to approximately 10 months
OS is defined as the time from randomization to death due to any cause. （Stage II） | Up to approximately 26 months

SECONDARY OUTCOMES:
Objective Response Rate (ORR) Per RECIST 1.1 as Assessed by Investigator （Stage I） | Up to approximately 26 months
Progression-free Survival (PFS) per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as Assessed by Investigator （Stage I） | Up to approximately 26 months
Disease Control Rate (DCR)up to approximately 26 months（Stage I） | up to approximately 26 months
Duration of Response (DOR) Per RECIST 1.1 as Assessed by Investigator （Stage I） | Up to approximately 26 months
Time to Progress(TTP) up to approximately 26 months（Stage I） | up to approximately 26 months
  The time from the date of the first medication to the date of the first recording of tumor progression (as measured according to THE RECIST v1.1 criteria, regardless of whether treatment is continued or not).
Overall survival (OS) up to approximately 26 months（Stage I） | up to approximately 26 months
Progression-free Survival (PFS) per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as Assessed by BIRC- and investigator（Stage II） | Up to approximately 26 months
Objective Response Rate (ORR) Per RECIST 1.1 as Assessed by BIRC- and investigator（Stage II） | Up to approximately 26 months
Disease Control Rate (DCR)Per RECIST 1.1 as Assessed by BIRC- and investigator（Stage II） | Up to approximately 26 months
Duration of Response (DOR) Per RECIST 1.1 as Assessed by BIRC- and investigator （Stage II） | Up to approximately 26 months
Time to Progress(TTP) up to approximately 26 months （Stage II） | up to approximately 26 months
  The time from the date of randomization to the date of the first recording of tumor progression (as measured according to THE RECIST v1.1 criteria, regardless of whether treatment is continued or not).
Incidence and severity of Participants Who Experience an Adverse Event (AE) as per NCI-CTC AE 5.0 （Stage II） | Up to approximately 26 months
Incidence and severity of Participants Who Experience a Serious AE (SAE) as per NCI-CTC AE 5.0（Stage II） | Up to approximately 26 months
Incidence and severity of Participants Who Experience an Immune-related AE (irAE) as per NCI-CTC AE 5.0（Stage II） | Up to approximately 26 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Feng J, Tang D, Wang J, Zhou Q, Peng J, Lou H, Sun Y, Cai Y, Chen H, Yang J, Liu P, Wang L, Zou J. SHR-1701, a Bifunctional Fusion Protein Targeting PD-L1 and TGFbeta, for Recurrent or Metastatic Cervical Cancer: A Clinical Expansion Cohort of a Phase I Study. Clin Cancer Res. 2022 Dec 15;28(24):5297-5305. doi: 10.1158/1078-0432.CCR-22-0346. PMID 35653122